CLINICAL TRIAL: NCT04953364
Title: Self-management for Amputee Rehabilitation Using Technology (SMART) Program: a Peer Supported mHealth Approach for Rehabilitation After Lower Limb Amputation
Brief Title: Self-Management for Amputee Rehabilitation Using Technology.
Acronym: SMART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, William C. Miller, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H20-03316
Record Dates: First submitted 2021-05-17; First posted 2021-07-08 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Behavior; Amputation; Lower Limb Amputation Above Knee (Injury); Lower Limb Amputation Below Knee (Injury); Lower Limb Amputation Knee
MeSH Terms: conditions — Behavior; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial (RCT)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMART (Experimental): The experimental group will receive access to SMART online platform (6 weeks). SMART includes mental and physical wellness, residual/prosthetic limb managements, use of a prosthesis and weekly peer-support calls or video call over Zoom, hosted by University of British Columbia, depends on participant's preference, promoting motivation and establishing goal setting and action planning. SMART will also allow asynchronous contact with trainers through a secure website.
  Interventions: Behavioral: SMART
- Control (Active Comparator): The control group will receive a care booklet and weekly contacts for 6 weeks.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: SMART — SMART includes mental and physical wellness, residual/prosthetic limb managements, use of a prosthesis and weekly peer-support calls or video call over Zoom, hosted by University of British Columbia, depends on participant's preference, promoting motivation and establishing goal setting and action planning. The tablet will also allow asynchronous contact with trainers through a secure website.
  Arms: SMART
Behavioral: Control — The control group will receive a care booklet and weekly contacts for 6 weeks.
  Arms: Control

SUMMARY:
Lower Limb Amputations (LLAs) are a substantial burden on the Canadian health services with nearly 50,000 cases reported between 2006 and 2011. To address the challenging nature of a LLA (e.g., decreased mobility, pain, depression), patients need to go through extensive rehabilitation programs. Effective self-management programs can help those with LLA to monitor their own condition and improve their quality of life. However, a lack of self-management programs, a limited healthcare budget, and a decrease in quality of services (e.g. shorter lengths of stay for inpatients and rapid movement to outpatient services) pose further challenges for patients with LLA. Self-management programs can be provided to clients through online mobile technologies (e.g., tablet) and offer accessible, low-cost, and potentially augmentative rehabilitation after discharge, in both urban and rural areas. To address these needs, an online educational and training platform for individuals with LLA called, Self-Management for Amputee Rehabilitation using Technology (SMART) was designed and developed. SMART focuses on LLA education, prosthetic limb management, and weekly support of peers. It is monitored by a trainer through a website. SMART will be evaluated in men and women with LLA aged 50 years and over, admitted to prosthetic rehabilitation throughout BC and ON. SMART has the potential to influence a client's post-LLA needs with direct (e.g., individual's health) and indirect (e.g., healthcare utilization) benefits. The purpose of this randomized controlled trial is to evaluate the effect of SMART in community dwelling older adults with unilateral, above or below, knee amputation.

DETAILED DESCRIPTION:
Importance: Amputation is a stressful experience which causes daily fluctuations in psychological and physical functioning and social interactions. Yearly, more than 7300 patients are admitted to hospitals nationwide for lower limb amputation (LLA), with the majority (86%) occurring in adults over 50. Consequences of LLA, such as a change in body image, mobility restrictions, and pain, may lead to depression, social isolation and decreased quality of life. Clients may lack coping strategies, educational resources, or access to rehabilitation services, especially for rural living Canadians. Online eHealth approaches, including the use of tablets, are considered effective approaches for delivering self-management programs, while addressing logistical barriers. Using a participatory action research approach, an eHealth platform for individuals with LLA called Self-Management for Amputee Rehabilitation using Technology (SMART) was co-designed and co-developed.

The investigators' goal is to determine the effectiveness and retention effect of SMART in community dwelling older adults (≥50yrs) with unilateral LLA, while documenting implementation factors. the hypothesis driving this investigation is that older adults with LLA who receive SMART intervention, compared with paper-based education as a control group, will have greater positive changes in confidence in their ambulation and walking capacity.

Methods: Using a Type 1 Effectiveness-Implementation Hybrid Design randomized controlled trial (RCT), the 6-week effectiveness and 4-week retention effect of SMART will be assessed on patient-relevant outcomes, and implementation. A volunteer sample of men and women, aged ≥50 years, with unilateral transtibial or transfemoral LLA, who started casting of their initial prosthetic limb, with command of English will be recruited from BC and ON. The sample will be randomly allocated to the experimental (SMART) (n=41) or control group (n=41), with a ratio of 1:1. Both groups will receive usual care, provided by their healthcare providers. The experimental group will receive a SMART enabled tablet for daily use (6 weeks). SMART includes mental and physical wellness, residual/prosthetic limb managements, use of a prosthesis and weekly peer-support calls or video call over Zoom, hosted by University of British Columbia, depends on participant's preference, promoting motivation and establishing goal setting and action planning. The tablet will also allow asynchronous contact with trainers through a secure website. The control group will receive a care booklet and weekly contacts. All data collection will be conducted using Zoom online platform, hosted by University of British Columbia. Confidence in ambulation will be measured by Ambulatory Self-Confidence Questionnaire (ASCQ) and Walking capacity will be assessed using the Timed Up and Go test (TUG)--these measures will be conducted under remote supervision via Zoom. Five elements of implementation will be assessed including, reach (target population), effectiveness (effects of SMART), adoption (by setting/staff), implementation (dose delivered and fidelity), and maintenance of the behavior (in target population and settings). Online one-on-one semi-structured interviews with 20 participants (SMART group) will be used to assess the participants' experience. The interviews will be conducted using Zoom video calls. Analyses: Outcomes will be disaggregated for sex and gender differences. Between- and within- group differences will be assessed by covariance analysis. Thematic analyses of qualitative data will explore participants' experience.

Noah Tregobov's role will be that of the research assistant. Elham Esfandiari will be coordinating most of the research as a graduate student.

William Miller is the PI and will oversee the overall execution of the project. All other team members will serve as resources for information, recruitment, research design, etc. but will not directly interact with participants.

ELIGIBILITY:
Inclusion Criteria:

* Has a unilateral LLA (transtibial or transfemoral) due to diabetes or vascular disease
* Received initial casting of their prosthesis within the past 2 years
* Be aged ≥ 50 years (85% of adults with LLA)
* Self-identifies as being able to speak and read English.
* Has access to computer or tablet and internet.
* Individuals living in British Columbia or Ontario, Canada.

Exclusion Criteria:

* Substantial health conditions (e.g., congestive heart failure, diagnosed dementia)
* Those anticipating further surgery (e.g. LLA revision) as identified by our study sites' physiatrists
* an inability to use a tablet (e.g. using hands for typing).

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2022-10-14 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
TUG, Timed Up and Go test | Ten weeks
  The patient stands up upon therapist's command: walks 3 meters, turns around, walks back to the chair and sits down.
ASCQ, the Ambulatory Self-Confidence Questionnaire | Ten weeks
  This questionnaire measures how confident you are in your ability to walk.
  Type of Administration:
  Self-Report.
  Response Scale:
  0 (not confident at all) - 10 (extremely confident)
  Scoring:
  Participants' total score is derived by calculating a mean score
  Interpretation:
  Higher scores = higher level of self-confidence regarding ambulation

SECONDARY OUTCOMES:
Self-Report Habit Index (SRHI) | Ten weeks
  12-item questionnaire based on the 7-point Likert scale with the range of total score between 0 to 84, which higher scores show the stronger habit strength
Physical Activity Identity (PAI) | Ten weeks
  Physical activity self-identification 7 point likert scale. Higher score = higher physical activity identification PAI items relate to how much the participant identifies with being physically active.
The Revised Amputee Body Image Scale (ABIS-R) | Ten weeks
  This questionnaire is designed to measure how you see and feel about your body image. It is not a test so there are no right or wrong answers. Please answer each item as carefully and as accurately as you can by placing the appropriate number beside each question as follows.
  Scale of 0, 1, 2. 0 = none of the time, 2 = most of the time High scores indicate high body image disturbance.
Center for Epidemiologic Studies Depression Scale (CES-D) | Ten weeks
  Below is a list of the ways you might have felt or behaved. Please tell me how often you have felt this way during the past week.
  20 items Scoring: 0, 1, 2, 3 representing "rarely" to "most of the time", respectively. The scoring of positive items is reversed. Possible range of scores is zero to 60, with the higher scores indicating the presence of more symptomatology.
Self-Report Habit Index (SRH) | Ten weeks
  Self report of limb cleaning tendencies
Activities Specific Balance Confidence (ABC) Scale | Ten weeks
  Assesses confidence in balance during different activities 16 items Each item is rated from 0% - 100% 100% indicates the participant is "completely confident" in the activity described in the item.
Residual limb pain, phantom pain, and non-painful phantom limb sensations | Ten weeks
  Residual limb pain, phantom pain, and non-painful phantom limb sensations
  Participants rate their pain on each of the 3 items. Scale of 1-10 Higher score means greater reported pain
Short Musculoskeletal Function Assessment (SMFA) | Ten weeks
  Items 1-34 of a questionnaire to assess the difficulty with daily activities and experiencing problems because of injury.
Euro Quality of Life | Ten weeks
  Five Level Instrument (EQ-5D-5L) assesses mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Tenacious goal pursuit (TGP) | Ten weeks
  Assesses tendency to persist and increase effort in pursuing goals facing obstacles
Action Planning Scale (AP) | Ten weeks
  Assesses whether people had formed a plan which links goal-directed behavior to environmental cues by indentifying when, where and how to act.
  We will specifically assess for 'exercising', 'skin monitoring', and 'cleaning the prosthesis'.
Self-Management Assessment Scale (SMASc) | Ten weeks
  Assesses five domains that are important for an effective self-management, including "knowledge, goals for future, daily routines, emotional adjustment, and social support".

CONTACTS AND LOCATIONS:
Overall Officials: William C Miller, PhD, Principal Investigator — The University of British Columbia
Locations (1):
- GF Strong Rehabilitation Centre, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Esfandiari E, Miller WC, King S, Payne M, Mortenson WB, Underwood H, MacKay C, Ashe MC. Protocol for a randomized controlled trial to assess the effect of Self-Management for Amputee Rehabilitation using Technology (SMART): An online self-management program for individuals with lower limb loss. PLoS One. 2023 Mar 23;18(3):e0278418. doi: 10.1371/journal.pone.0278418. eCollection 2023. PMID 36952517